CLINICAL TRIAL: NCT06425666
Title: European Prospective Multicentre Trial Comparing Cataract Surgery With Triple-DMEK in Patients With Cataract and Fuchs Endothelial Corneal Dystrophy (ETCF-trial)
Brief Title: Trial Comparing Cataract Surgery With Triple-DMEK in Patients With Cataract and Fuchs Endothelial Corneal Dystrophy
Acronym: ETCF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: The Clinical Trials Centre Cologne (Other); ESCRS (European Society of Cataract and Refractive Surgeons) (Unknown)
Responsible Party: Principal Investigator, Björn Bachmann, Clinical Professor, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-5135; ORG-100006227 (Other: ESCRS (European society of Cataract and Refractive Surgeons))
Record Dates: First submitted 2024-05-02; First posted 2024-05-22 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-11

CONDITIONS: Cataract Surgery; Cataract and Fuchs Endothelial Corneal Dystrophy
Keywords: Fuchs´ Endothelial Corneal Dystrophy Krachmer grade 3 and 4; nuclear cataract; Nuclear opalescence (NO) grades 2; Nuclear opalescence (NO) grades 3; Central corneal thickness
MeSH Terms: conditions — Cataract; Fuchs' Endothelial Dystrophy | interventions — Cataract Extraction; Control Groups

STUDY DESIGN:
Intervention Model Description: The trial will be a prospective, randomised, controlled, European, multicentre, open clinical trial in which patients with FECD and cataract will receive either cataract surgery without DMEK (intervention goup/arm 1) or triple-DMEK (DMEK in combination with cataract surgery; control group/arm 2).
  (Protocol V02_0_TC page 37)
Masking Description: After screening and enrollement subjects will be randomly allocated to the trial groups (cataract surgery versus triple-DMEK, allocation rate 1:1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental intervention /arm 1 (Experimental): After randomisation the investigational therapy (arm 1), patients undergo a cataract surgery with preservation of the diseased endothelial cells. The cataract surgery will take approximately 10-20 minutes.
  The follow-up period after surgery will be 22 weeks ± 14 days.
  Interventions: Procedure: Intervention group /arm 1 (Cataract surgery alone)
- Control intervention /arm2 (Other): After randomisation, patients in the comparator therapy (arm 2) undergo triple-DMEK which is a cataract surgery combined with DMEK (removal of the diseased endothelial cells followed by transplantation of a healthy endothelial cell layer).
  Triple-DMEK takes approximately 5-10 minutes longer than cataract surgery. The follow-up period after surgery will be 22 weeks ± 14 days.
  Interventions: Procedure: Control group /arm 2: Corneal transplantation as Descemet Membrane Endothelial Keratoplasty (DMEK) in combination with cataract surgery (triple-DMEK)

INTERVENTIONS:
Procedure: Intervention group /arm 1 (Cataract surgery alone) — Cataract surgery (arm 1) is performed using a small incision technique. The tunnel is used both for cataract surgery and for implantation of the DMEK graft (arm 2). The centres confirmed that the main incision will be localized between 11 and 12 o'clock and will have a width of 2.4 to 2.8 mm. A tunnel suture will only be placed if there is leakage from the incisions. If cataract surgery alone (arm 1) is performed, a thin dispersive viscoelastic is applied to the endothelium for protection before phacoemulsification. A hydrophobic acrylic monofocal IOL will be implanted into the bag. The centers confirmed that Barret Universal II formula is the standard IOL calculation formula for both groups and for all axial lengths.
  Arms: Experimental intervention /arm 1
Procedure: Control group /arm 2: Corneal transplantation as Descemet Membrane Endothelial Keratoplasty (DMEK) in combination with cataract surgery (triple-DMEK) — After cataract surgery DMEK is continued using the surgeon's standard technique for graft implantation and unfolding in triple-DMEK. In all cases the graft will be implanted using the same main incision as for IOL implantation. Once the DMEK graft is unrolled and attached to the posterior corneal stroma the complete anterior chamber will be filled with SF6 20%.
  Arms: Control intervention /arm2

SUMMARY:
The purpose of the study is to investigate whether there is a difference in BCVA in patients who receive one of the following two surgeries: intervention group (arm 1) cataract surgery alone and control group (arm 2) cataract surgery combined with removal of the diseased endothelial cells and the attached Descemet's membrane followed by transplantation of a healthy endothelial cell layer with attached Descemet's membrane ("triple-DMEK" group; comparator therapy).

The secondary objectives are to compare the two surgical methods with regard to other visual functions and optical as well as morphological differences, to safety, to quality of life, and to safety.

DETAILED DESCRIPTION:
After signing the informed consent, patients are screened for eligibility for the trial regarding in- and exclusion criteria.

Different tests will be performed like ocular examination including slit lamp examination, fundus examination, IOP measurement, BCVA, Pentacam imaging, and Macular-OCT, vital signs. In addition, women below age of 60 have to perform a urine pregnancy test. Once all inclusion criteria and none of the exclusion criteria are met, the patient will be enrolled into the trial and will receive a subject-ID.

The Baseline Visit can take place up to 7 days after enrolment of the subject into the clinical trial. At the Baseline Visit a photograph of the cornea in retroillumination will be taken (can be taken either at Screening & Enrolment Visit or at Baseline Visit) and uploaded into the eCRF for central grading by CORIC.

In addition, subjects have to complete vision related quality of life questionnaires and changes in relevant medical history/concomitant diseases as well as concomitant medications have to be documented.

Furthermore, a contrast sensitivity test and an optical quality test (if device available) will be peformed.

After all investigations are completed, the subject will be randomised via the central 24-7 Internetrandomisation service ALEA and distributed to the respective treatment groups.

Intervention (surgery):

On that day and before starting intervention all women below 60 years undergo a pregnancy test and changes in relevant medical history/concomitant diseases have to be documented. In arm 1 (intervention group) patients undergo exclusively cataract surgery, in arm 2 (control group) patients undergo triple-DMEK, i.e. cataract surgery and DMEK.

The immediate follow-up appointments for clinical examinations are, as per standard of care, at the discretion of the respective trial centres treating physician.

The Post-operative Visit will take place 22 weeks ± 14 days after the surgical intervention. During the Post-operative Visit an ocular examination including slit lamp examination, fundus examination, IOP measurement, BCVA, Pentacam imaging, contrast sensivity test, an optical quality test (if device available), and Macular-OCT will be performed. In addition, vital signs will be taken and subjects have to complete the vision related quality-of-life questionnaires again. Concomitant medications and AEs/SAEs have to be documented.

The duration of the clinical trial for every individual subject will be up to 29 weeks (time from Screening & Enrolment Visit to Post-operative Visit).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with FECD and nuclear cataract in study eye
2. Male and female patients ≥18 years of age
3. Subject must be able to understand and read the national language.
4. Written informed consent prior to any study-related procedures
5. Nuclear opalescence (NO) grades 2 and 3 according to the lens opacities classification system III (LOCS III)
6. Krachmer grade (3 [2-5 mm diameter area with confluent guttae]; 4 [ > 5 mm diameter area with confluent guttae] without edema identified by slit lamp examination)
7. Central corneal thickness (CCT) measured with Pentacam below 620 µm between 8:00 am and 01:00 pm
8. BCVA logMAR < 0,7 and > 0,1
9. No previous cataract surgery or triple-DMEK on the opposite side
10. Pentacam quality specification: "OK"
11. For women below age of 60 negative urine pregnancy test

Exclusion Criteria:

1. Patients with ocular and/or systemic comorbidity affecting vision or clinically proven anterior and/or posterior segment disease other than FECD and cataract (exclusion of macular disease or edema by OCT)
2. Iris synechiae, pupil diameter <6 mm after dilatation, pseudoexfoliation syndrome, subluxated lens, previous history of ocular trauma/surgery or inflammatory disease
3. Subjective diurnal changes in visual acuity with worse visual acuity in the morning
4. Corneal (epithelial) edema visible at slit lamp examination
5. Preoperative anterior chamber depth below 2 mm
6. Participation in other interventional trials parallel or within the last 4 weeks
7. Systemic use of Alpha-1-Adrenozeptor-Antagonists, immunosuppressive therapy or chemotherapy
8. Pregnant women and nursing mothers
9. Persons with any kind of dependency on the principal investigator or employed by the sponsor or principal investigator
10. Legally incapacitated persons
11. Persons held in an institution by legal or official order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
BCVA 22 | 22 weeks +/- 14 days after surgery
  Best corrected visual acuity (BCVA) is messured with EDTRS-charts (transformed to logMAR)

SECONDARY OUTCOMES:
Change in visual acuity (BCVA) | Baseline (pre-op) and 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: ETDRS-charts (transformed to logMAR); Analysis metric (participant level): Difference value at follow-up- baseline value Method of aggregation (summary measure for each study group): Mean difference
Contrast sensitivity | 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Total score of Freiburg Vision Test "FrACT"; Analysis metric (participant level): Value Method of aggregation (summary measure for each study group): Mean
Change in contrast sensitivity | 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Total score of Freiburg Vision Test "FrACT"; Analysis metric (participant level): Difference Value at follow-up-baseline value; Method of aggregation (summary measure for each study group): Mean difference
Optical quality measured by HD-analyzer | 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Total score of objective scattering index (OSI); Analysis metric (participant level): Value Method of aggregation (summary measure for each study group): Mean
Change in optical quality measured by HD-analyzer | 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Total score of objective scattering index (OSI); Analysis metric (participant level): Difference value at follow-up- baseline value Method of aggregation (summary measure for each study group): Mean difference
Optical quality measured by HD-analyzer | 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Total score of Modulation transfer function (MTF) cut-off; Analysis metric (participant level): value Method of aggregation (summary measure for each study group): Mean
Change in optical quality measured by HD-analyzer | 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Total score of Modulation transfer function (MTF) cut-off; Analysis metric (participant level): Difference value at follow-up - baseline value Method of aggregation (summary measure for each study group): Mean difference
Optical quality measured by HD-analyzer | 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Total score of Strehl ratio; Analysis metric (participant level): Value Method of aggregation (summary measure for each study group): Mean
Change in Optical quality measured by HD-analyzer | 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Total score of Strehl ratio; Analysis metric (participant level): Difference value at follow-up- baseline value Method of aggregation (summary measure for each study group): Mean difference
Refractive accuracy:spherical equivalent | 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Deviation from target refraction from IOL calculation [D], Analysis metric (participant level): Value Method of aggregation (summary measure for each study group): Mean numerical prediction error (ME) and Mean absolute prediction error (MAE)
Corneal topography/ tomography parameters | 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Corneal densitometry (grayscale unit GSU) (anterior, central, posterior and total layer) Analysis metric (participant level): Value; Method of aggregation (summary measure for each study group): Mean
Change in corneal topography/tomography parameters | At baseline and 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Corneal densitometry (grayscale unit GSU) (anterior, central, posterior and total layer); Analysis metric (participant level): Difference value at follow-up - baseline value; Method of aggregation (summary measure for each study group): Mean difference
Central corneal thickness (CCT) | At baseline and 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: CCT measured by Pentacam [μm]; Analysis metric (participant level): Value; Method of aggregation (summary measure for each study group): Mean
Change in central corneal thickness (CCT) | At baseline and 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: CCT measured by Pentacam [μm]; Analysis metric (participant level): Difference value at follow-up - baseline value Method of aggregation (summary measure for each study group): Mean difference
Quality of life | 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Catquest-9SF (all centers) and V-Fuchs (Germany only); Analysis metric (participant level): Total score [no dimension]; Method of aggregation (summary measure for each study group): Mean
Change in quality of life | At baseline and at 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Catquest-9SF (all centers) and V-Fuchs (Germany only); Analysis metric (participant level): Difference total score at follow-up- baseline total score; Method of aggregation (summary measure for each study group): Mean difference
Change in central retinal thickness | At baseline and at 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Measured by OCT Analysis metric (participant level): Difference value at follow-up- baseline value; Method of aggregation (summary measure for each study group): Mean difference
Change in intraocular pressure (IOP) | At baseline and at 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: IOP [mmHg] Analysis metric (participant level): Difference value at follow-up - baseline value Method of aggregation (summary measure for each study group): Mean difference
Additional ocular surgeries | At baseline and at 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Per patient anamnesis Analysis metric (participant level): Value (yes/no) Method of aggregation (summary measure for each study group): Proportion
Endothelial decompensation with indication for endothelial keratoplasty (either planned or already performed) | 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: Per patient anamnesis (decision made by treating ophthalmologist; incl. ophthalmologist outside the study team) Analysis metric (participant level): Value [yes/no] Method of aggregation (summary measure for each study group): Proportion
Cystoid macular edema | 22 weeks +/- 14 days after initial surgery
  Specific measurement variable: CME visualized by OCT Analysis metric (participant level): Value [yes/no] Method of aggregation (summary measure for each study group): Proportion

CONTACTS AND LOCATIONS:
Overall Officials: Björn Bachmann, Prof., Principal Investigator — University Hospital Cologne
Locations (4):
- Department of Ophthalmology, Aarhus University Hospital, Aarhus N, Central Jutland, Denmark
- Klinik für Ophthalmologie des Universitätsklinikums Köln, Cologne, North Rhine-Westphalia, Germany
- Radboud-Universität Nijmegen, Nijmegen, Gelderland, Netherlands
- Instituto de microcirugía ocular; Departamento de Cornea y Cirugia Refractiva, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No